CLINICAL TRIAL: NCT00502762
Title: Salvage Treatment With Topotecan in Patients With Irinotecan-Refractory Small Cell Lung Cancer
Brief Title: Topotecan for Irinotecan-Refractory SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gachon University Gil Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMO-LU-51
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2008-03-12 (Estimated); Status verified 2008-03

CONDITIONS: Lung Cancer; Refractory to Chemotherapy
Keywords: small-cell lung cancer; refractory; topotecan
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: topotecan

SUMMARY:
Although the efficacy of topotecan as second-line chemotherapy for SCLC has been consistently demonstrated in phase II/III clinical trials, the choice of irinotecan as first-line therapy prevented use of the evidence-based option.

This pilot study will be conducted to determine the activity and safety of topotecan in SCLC patients refractory to first-line therapy with irinotecan and platinum.

DETAILED DESCRIPTION:
Current commonly used second-line approaches for SCLC include re-induction with first-line therapy for chemosensitive disease, or single-agent topotecan. Although the efficacy of topotecan as second-line chemotherapy for SCLC has been consistently demonstrated in a number of clinical studies, the choice of irinotecan as first-line therapy prevented use of the evidence-based option such as topotecan. Topotecan and irinotecan are cytotoxic agents that inhibit same intracellular pathway, namely topoisomerase I, which is an enzyme involved in DNA replication and RNA transcription.

Although their mechanism of action is similar, the preclinical and clinical data of these two drugs have some notable differences. Topotecan and irinotecan have different spectra of antitumor activity in various models of human cancer. Clinical data support that these agents may have different spectra of activity. The differences in antitumor activities may also reflect different mechanisms of resistance. Furthermore, topotecan and irinotecan have different limiting toxicities (myelosuppression and diarrhea, respectively).

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven SCLC
* refractory to prior irinotecan-based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* age between 18 and 75 years
* no active brain or leptomeningeal metastases
* adequate hematologic, hepatic and renal functions
* at least one measurable lesion(s)

Exclusion Criteria:

* pregnant or lactating women
* patients with active infection
* extensive radiotherapy within the previous 4 weeks
* previous other malignancies with the exception of adequately treated non-melanoma skin cancer or in situ cervical cancer
* any severe comorbid illness
* a known history of anaphylaxis of any origin
* history of severe adverse events to the drug used in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-09; Study Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
Response rate

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Eun Kyung Cho, MD, Principal Investigator — Gachon University Gil Medical Center, Incheon, Korea
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea